CLINICAL TRIAL: NCT01485822
Title: A Multicenter Study of the Pigmentation in the Trabecular Meshwork After Two Years of Treatment With TRAVATAN 0.004% Ophthalmic Solution
Status: Terminated | Type: Observational
Why Stopped: Study objectives met
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: C-01-78
Record Dates: First submitted 2011-12-01; First posted 2011-12-06 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Open-angle Glaucoma
Keywords: Glaucoma; Travatan; Trabeculectomy
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Travoprost; Ophthalmic Solutions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TRAVATAN: As prescribed by physician for the treatment of open-angle glaucoma and dosed for at least two years
  Interventions: Procedure: Trabecular Meshwork Tissue Collection; Drug: Travoprost 0.004% ophthalmic solution
- Treatment Naive: No prior exposure (or less than 1 month) to any topical, ocular prostaglandin analogue
  Interventions: Procedure: Trabecular Meshwork Tissue Collection

INTERVENTIONS:
Procedure: Trabecular Meshwork Tissue Collection — A minimum of two punches were used to remove tissue to form a sclerostomy. Tissue removed by the punch was collected for analysis. Alternatively, the tissue was collected by block excision of the meshwork with scissors at the time of sclerostomy.
Drug: Travoprost 0.004% ophthalmic solution
  Other Names: TRAVATAN Z; TRAVATAN
  Groups: TRAVATAN

SUMMARY:
The purpose of this study was to assess the pigmentation in the trabecular meshwork of patients who had been treated for at least 2 years with TRAVATAN compared with patients without exposure (or less than 1 month) to a prostaglandin analogue (PGA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma without pseudoexfoliation or pigment dispersion component;
* Either two or more years of dosing with Travatan, or no prior exposure (less than 1 month) to a topical ocular prostaglandin;
* Requires a trabeculectomy;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Pseudoexfoliation or pigment dispersion;
* History of chronic or recurrent severe inflammatory eye disease;
* History of or current ocular infection or ocular inflammation within the past 3 months in either eye;
* Greater than one month but less than two years of exposure to TRAVATAN;
* Pregnant, breast-feeding, not using highly effective birth control;
* Other protocol-defined exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were identified and enrolled from 9 study centers in the US and 1 in Spain.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2004-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Melanin Granule Count | Day 1
  A trabecular meshwork tissue sample was collected by the investigator. The number of pigment granules was counted for three separate microscopic fields of view. Mean melanin granule count was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Landry, PhD, Study Director — Alcon Research